CLINICAL TRIAL: NCT06051825
Title: Diagnostic Importance of the Circulating C-reactive Protein in Blood and Saliva in Acute Appendicitis in Pediatric Patients
Brief Title: Diagnostic Importance of the C-reactive Protein From Blood and Saliva in Children With Acute Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Klaudio Pjer Milunovic, principal investigator, University Hospital of Split
Other Study IDs: CHCSplit
Record Dates: First submitted 2023-09-07; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acute appendicitis: Patients with acute appendicitis, after surgery and with pathohistological confirmation
  Interventions: Diagnostic Test: Blood specimen collection for C-reactive protein (CRP) and WBC (white blood cells). Saliva specimen collection for analysis of CRP levels
- Patients without acute appendicitis: Patients without acute appendicitis, after laboratory, clinical and/or radiological exclusion of acute admittance
  Interventions: Diagnostic Test: Blood specimen collection for C-reactive protein (CRP) and WBC (white blood cells). Saliva specimen collection for analysis of CRP levels

INTERVENTIONS:
Diagnostic Test: Blood specimen collection for C-reactive protein (CRP) and WBC (white blood cells). Saliva specimen collection for analysis of CRP levels — Blood analysis of CRP and WBC levels Saliva analysis of CRP levels

SUMMARY:
Diagnosing acute appendicitis in children is still a challenge even for experienced clinicians. Failure to recognize this acute condition can result in perforation, with consequent peritonitis, or misdiagnosis can result in negative appendectomies. C-reactive protein in blood can be elavated in children with acute appendicitis. The aim of this research is to compare the diagnostic value of C-reactive protein from the blood and saliva of children with acute appendicitis and to prove wheter the analysis of biomarker from saliva as a minimally invasive procedure can be sufficient for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* children with age from 5 to 17 with acute abdominal pain
* children with clinical signs of appendicitis

Exclusion Criteria:

* previous diagnosis of chronic and/or malignant disease
* children wich had previous abdominal surgery
* pregnancy

Ages: 5 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Patients from 5 to 17 years of age, presenting with acute abdominal pain consistent with diagnosis of acute appendicitis, to Emergency Surgery Department at the University Hospital Split
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Level of CRP in blood | 72 hours
  Levels of CRP in blood as measured by ELISA test

SECONDARY OUTCOMES:
Level of CRP in saliva | 72 hours
  Levels of CRP in saliva as measured by ELISA test

CONTACTS AND LOCATIONS:
Overall Officials: Zenon Pogorelić, PhD.Prof, Principal Investigator — University Hospital of Split

IPD SHARING:
Plan to Share IPD: No